CLINICAL TRIAL: NCT04861402
Title: Non-Invasive Intracranial Pressure in COVID-19 Individuals
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Sens4care (Industry)
Responsible Party: Principal Investigator, Gisele Sampaio Silva, Gisele Sampaio Silva, Federal University of São Paulo
Other Study IDs: 31589920.7.1001.5505
Record Dates: First submitted 2021-04-25; First posted 2021-04-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Pressure
Keywords: Neurocritical care, Infectious Disease Medicine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Non-intubated COVID-19 group: Men and women (not pregnant) Older than 18 years old Diagnosis of COVID-19 confirmed by Reverse Transcription Polymerase Chain Reaction (RT-PCR) Subjects intubated Time between admission and study inclusion ≤ 72h Non-intubated during the monitoring carried out in the study Time between onset symptoms and study inclusion ≤ 14 days No neurological acute disease No cutaneous injury in the head to impossibility the ICP monitoring No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously.
  Interventions: Device: The ICP monitoring will be performed in a non-invasive method developed by Brain4Care
- Intubated COVID-19 group: Men and women (not pregnant) Older than 18 years old Diagnosis of COVID-19 confirmed by Reverse Transcription Polymerase Chain Reaction (RT-PCR) Subjects intubated Time between admission and study inclusion ≤ 72h For intubated group time between IUC admission and study inclusion ≤ 72h Time between onset symptoms and study inclusion ≤ 14 days No neurological acute disease No cutaneous injury in the head to impossibility the ICP monitoring No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously.
  Interventions: Device: The ICP monitoring will be performed in a non-invasive method developed by Brain4Care
- Health control group: Men and women (not pregnant) Older than 18 years old No cutaneous injury in the head to impossibility the ICP monitoring No symptoms of COVID-19 on the last 15 days
  • For healthy group: No previous neurological disease No chronic disease as Diabetes Mellitus Type 2, Chronic Obstructive Pulmonary Disease (COPD), Heart Failure, hypertension or Chronic Kidney Disease (CKD) No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously.
  Interventions: Device: The ICP monitoring will be performed in a non-invasive method developed by Brain4Care
- Non-COVID-19 and non-neurological disease intubated group: Men and women (not pregnant) Older than 18 years old No cutaneous injury in the head to impossibility the ICP monitoring
  • For intubated group: ICF signed by the participant or his/her legal representative* Intubated patients for others causes than COVID-19 or neurological diseases IUC admission and study inclusion ≤ 72h No symptoms of COVID-19 on the last 15 days No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously.
  Interventions: Device: The ICP monitoring will be performed in a non-invasive method developed by Brain4Care

INTERVENTIONS:
Device: The ICP monitoring will be performed in a non-invasive method developed by Brain4Care — The ICP monitoring will be performed in a non-invasive way through the cranial deformation method developed by Brain4Care Inc.
  The selected patients will be monitored until 1h/day for 7 sequential days or even discharge. The clinical outcomes such as ventilatory status will be noted (if the subject is under oxygen supplementation, using non-invasive mechanical ventilation or intubated), the ventilatory parameters during the monitorization will be analyzed in the intubated group (or those from a non-intubated group who was intubated during the seven days of hospitalization) including IFO2, CV, PEEP, driving pressure, and pressure plate as well as ventilatory asynchronies. Some changes in ventilatory parameters during monitorization will be noted. These procedures will be applied to all groups, excepted to the healthy group. This last group will be monitored only once for 30 minutes at the Federal University of São Carlos (UFSCar).
  Other Names: The presence of spontaneous microembolization will be assessed by means of non-invasive monitoring by transcranial doppler

SUMMARY:
The use of non-invasive intracranial pressure monitoring, including intracranial pressure pulse morphology in patients with COVID-19, could calculate possible components associated with the presence of neurological symptoms in these patients, in addition to being a tool with the potential to monitor the repercussion of MV at cerebral compliance patient patients. In addition, it is likely that patients with COVID-19 also have cerebral embolization more frequently than healthy patients, which is justified by transcranial doppler ultrasound assessment. The aim of the study is to monitor this brain pressure using a non-invasive method of monitoring, with a helmet-like system in place, for 1 hour for 7 consecutive days. There will be no associated invasive procedure of any kind. Monitoring will be done by the criteria themselves, no place where the patient and the mandatory volunteer. Another objective is to capture signs of microembolisms (small strokes that have not yet manifested) by performing a doppler ultrasound on the head with a helmet also for 1 hour, in a single evaluation.

The study population will include inpatients with COVID-19 infection. The control group will be in patients who do not have Covid-19. The control group will consist of people with similar characteristics and who have not recovered. Patients who meet the inclusion criteria incorporated into the monitoring with a non-invasive intracranial pressure device for 1 hour during hospitalization (Brain4Care® device approved by ANVISA), being monitored for up to seven days, in addition to monitoring for 1 hour with a transcranial doppler ultrasound helmet DWL® in a single assessment. There will be no invasive procedures or other equipment used without due knowledge by Organs competent bodies. It does not collect collection or retention of any biological material.

DETAILED DESCRIPTION:
INTRODUCTION: The Coronavirus Disease 2019 (COVID-19) is an infectious disease transmitted one person to another mainly from cough and sneeze aerosols as well as from contaminated surfaces. The most common respiratory symptoms are dry cough, fever, and dyspnea, but the Severe Respiratory Acute Syndrome (SARS) can be installed increasing disease´s mortality. In addition, neurological symptoms have been described according the increase of severity and age. Changes of intracranial pressure (ICP) can partially explain the Central Nervous System (CNS) impairment due to COVID-19. The ICP waveform can bring relevant information about intracranial compliance, and, nowadays, it can be measured by non-invasive technology. Clinically, non-invasive ICP waveform assessment would help to understand the repercussion of Invasive Mechanical Ventilation (IMV) on CNS in COVID-19 persons. AIMS: This study aims to evaluate the ICP waveform in intubated and non-intubated COVID-19 persons. Furthermore, the association between ICP and IMV parameters, level of sedation, heart rate variability, neurological symptoms, neuroimage, and final discharge will be investigated. . METHODS: At least 30 COVID-19 individuals will be included within 72h from admission and 14 days from symptoms onset. They will be divided into two groups: non-intubated (n=15) and intubated, paired with non-COVID-19 ones (non-intubated and intubated non-COVID-19 groups, respectively). The non-invasive ICP monitoring will be daily performed for 7 consecutive days. The Brain4Care's device and Analytic System will be used to assess the three pulse peaks (P1, 2 and 3) at the ICP waveform. The following variables will be investigated: P1 and P2 amplitude, P2/P1 ratio, time to peak and time percentage of P2 higher than P1. For statistics, all variables will be tested as to their normal or non-normal distribution through appropriate statical analyzes. For basic demographic and clinical variables, descriptive data analysis will be used. The repetitive measurement Anova will be used for ICP outcomes throughout the days. Pearson's or Spearman´s correlations will be applied according to data distribution.

ELIGIBILITY:
Inclusion Criteria:

For COVID-19 group:

* Men and women (not pregnant) Older than 18 years old Diagnosis of COVID-19 confirmed by Reverse Transcription Polymerase Chain Reaction (RT-PCR) Subjects intubated or non-intubated Time between admission and study inclusion ≤ 72h For intubated group time between IUC admission and study inclusion ≤ 72h Time between onset symptoms and study inclusion ≤ 14 days No neurological acute disease No cutaneous injury in the head to impossibility the ICP monitoring ICF signed by the participant or his/her legal representative*

No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously. Subjects intubated or non-intubated For intubated group time between IUC admission and study inclusion ≤ 72h Time between admission and study inclusion ≤ 72h Time between onset symptoms and study inclusion ≤14 days No neurological acute disease

For Controls Group:

Men and women (not pregnant) Older than 18 years old No cutaneous injury in the head to impossibility the ICP monitoring • For intubated group: ICF signed by the participant or his/her legal representative* Intubated patients for others causes than COVID-19 or neurological diseases IUC admission and study inclusion ≤ 72h No symptoms of COVID-19 on the last 15 days

• For healthy group: No previous neurological disease No chronic disease as Diabetes Mellitus Type 2, Chronic Obstructive Pulmonary Disease (COPD), Heart Failure, hypertension or Chronic Kidney Disease (CKD)

No cutaneous injury in the head to impossibility the monitoring with the transcranial doppler helmet Patients who have not been submitted to decompressive craniectomy previously.

IUC admission and study inclusion ≤ 72h No neurological diseases

Exclusion Criteria:

* It will be excluded those who asked to stop their participation, and those with problems in acquiring ICP data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a multicenter longitudinal study of 4 centers in Brazil: Hospital of São Paulo (Federal University of São Paulo), Benemérita Portuguese Charity Association, São Paulo-SP, ESHO Hospital Services Company AS, São Paulo, SP and Federal University of São Carlos, São Carlos-SP, from June to December of 2020. This will follow Helsinki recommendations for human protocols. This study was approved by Federal University of São Paulo's Human Research Ethics Committee (process number 4,050,985). The patients who completed the inclusion criteria (table 1) will be invited to participate, and they will receive an Informed Consent Form (ICF).
  At least 60 subjects will be included, and they will be equally divided into 4 groups.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
ICP pulse waveform | 01/06/2021
  To evaluate the ICP pulse waveform in patients with COVID-19 non-intubated compared to healthy subjects.
ICP pulse waveform 2 | 01/06/2021
  To evaluate the ICP pulse waveform in intubated patients with COVID-19 compared to intubated subjects with other diagnoses except COVID-19.
spontaneous microemboli | 01/06/2021
  To evaluate the spontaneous microemboli presence with TCD in those subjects who received the ICP monitoring.

SECONDARY OUTCOMES:
Secondary Outcome | 01/06/21
  To correlate the ICP pulse waveform and the presence of neurological symptoms on hospital admission in the non-intubated COVID-19 group
Secondary Outcome 1 | 01/06/2021
  To correlate the ICP pulse waveform and the emergence of neurological symptoms during the admission in the non-intubated COVID-19 group
Secondary Outcome 2 | 01/06/2021
  To correlate the ICP pulse waveform and the necessity of intubation during hospitalization time in the non-intubated COVID-19 group
Secondary Outcome 3 | 01/06/2021
  To correlate the ICP pulse waveform and the Heart Rate Variability in the non-intubated COVID-19 group
Secondary Outcome 4 | 01/06/2021
  To correlate the ICP pulse waveform and neuroimaging when available in the non-intubated COVID-19 group
Secondary Outcome 5 | 01/06/2021
  To correlate the ICP pulse waveform and the outcome on discharge in the non-intubated COVID-19 group
Secondary Outcome 6 | 01/06/2021
  To correlate the ICP pulse waveform to ventilatory parameters (inspired fraction of oxygen [IFO2], PEEP, Current Volum [CV] and driving pressure) in the intubated COVID-19 group
Secondary Outcome 7 | 01/06/2021
  To correlate the ICP pulse waveform to sedation used in the intubated COVID-19 group
Secondary Outcome 8 | 01/06/2021
  To correlate the ICP pulse waveform to HRV in the intubated COVID-19 group
Secondary Outcome 9 | 01/06/2021
  To correlate the ICP pulse waveform and the neurological symptoms on hospital admission in the intubated COVID-19 group
Secondary Outcome 10 | 01/06/2021
  To correlate the ICP pulse waveform and the outcome at hospital discharge in the intubated COVID-19 group
Secondary Outcome 11 | 01/06/2021
  To correlate the ICP pulse waveform and to neuroimaging when available in the intubated COVID-19 group

CONTACTS AND LOCATIONS:
Overall Officials: GISELE GS SILVA, SAMPAIO, Principal Investigator — Uf SAO PAULO
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
There isn't defined a plan to make individual participant data (IPD) available to other researchers yet.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: for research
Access Criteria: for research

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhou P, Yang XL, Wang XG, Hu B, Zhang L, Zhang W, Si HR, Zhu Y, Li B, Huang CL, Chen HD, Chen J, Luo Y, Guo H, Jiang RD, Liu MQ, Chen Y, Shen XR, Wang X, Zheng XS, Zhao K, Chen QJ, Deng F, Liu LL, Yan B, Zhan FX, Wang YY, Xiao GF, Shi ZL. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020 Mar;579(7798):270-273. doi: 10.1038/s41586-020-2012-7. Epub 2020 Feb 3. PMID 32015507
- [Background] Jin Y, Yang H, Ji W, Wu W, Chen S, Zhang W, Duan G. Virology, Epidemiology, Pathogenesis, and Control of COVID-19. Viruses. 2020 Mar 27;12(4):372. doi: 10.3390/v12040372. PMID 32230900
- [Background] Su S, Wong G, Shi W, Liu J, Lai ACK, Zhou J, Liu W, Bi Y, Gao GF. Epidemiology, Genetic Recombination, and Pathogenesis of Coronaviruses. Trends Microbiol. 2016 Jun;24(6):490-502. doi: 10.1016/j.tim.2016.03.003. Epub 2016 Mar 21. PMID 27012512
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Donoghue M, Hsieh F, Baronas E, Godbout K, Gosselin M, Stagliano N, Donovan M, Woolf B, Robison K, Jeyaseelan R, Breitbart RE, Acton S. A novel angiotensin-converting enzyme-related carboxypeptidase (ACE2) converts angiotensin I to angiotensin 1-9. Circ Res. 2000 Sep 1;87(5):E1-9. doi: 10.1161/01.res.87.5.e1. PMID 10969042
- [Background] Ye M, Ren Y, Lv T. Encephalitis as a clinical manifestation of COVID-19. Brain Behav Immun. 2020 Aug;88:945-946. doi: 10.1016/j.bbi.2020.04.017. Epub 2020 Apr 10. No abstract available. PMID 32283294
- [Background] Paniz-Mondolfi A, Bryce C, Grimes Z, Gordon RE, Reidy J, Lednicky J, Sordillo EM, Fowkes M. Central nervous system involvement by severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). J Med Virol. 2020 Jul;92(7):699-702. doi: 10.1002/jmv.25915. PMID 32314810